CLINICAL TRIAL: NCT00044772
Title: A Double-blind, Placebo-controlled, Parallel-group Comparison of Venlafaxine Extended-release Capsules and Paroxetine in Outpatients With Panic Disorder
Brief Title: Study Evaluating Venlafaxine ER in Patients With Panic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0600B5-399
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Panic Disorder
Keywords: Panic; Disorder
MeSH Terms: conditions — Panic Disorder; Disease

INTERVENTIONS:
Drug: Venlafaxine ER

SUMMARY:
The primary objective is to determine the efficacy, safety, and tolerability of venlafaxine extended release (ER) capsules in the treatment of outpatients with panic disorder (PD) in comparison to those of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for PD (with or without agoraphobia) for at least 3 months before study day 1
* Have sufficient symptoms to require anxiolytic drug therapy
* Have a score ≥4 on the Clinical Global Impressions Scale (CGI) severity of illness item at screening and baseline

Exclusion Criteria:

* Known hypersensitivity to venlafaxine (IR or ER), related compounds, or paroxetine
* History or presence of any clinically important hepatic, renal, or other medical disease that might compromise the study or be detrimental to the patient (eg, clinically important cardiac arrhythmia, unstable diabetes, carcinoma [except basal cell epithelioma], uncontrolled hypertension)
* Clinically important abnormality on screening physical examination, vital signs, electrocardiogram (ECG), laboratory tests or urine drug screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2001-11; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer